CLINICAL TRIAL: NCT03584945
Title: Task Control Circuit Targets for Obsessive Compulsive Behaviors in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Columbia University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kate D. Fitzgerald, Professor, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00144074; 1R01MH114958-01A1 (NIH); R01MH115024-01A1 (NIH)
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Obsessive-compulsive Disorders and Symptoms in Children
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Children ages 6-14 with OCD, obsessive compulsive symptoms, or healthy controls
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Obsessive Compulsive Disorder (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Subclinical Obsessive-Compulsive symptoms (OCS) (Other)
  Interventions: Other: Community Referral as appropriate
- Healthy Control (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The treatment team will offer a course of up to 12 cognitive behavioral therapy (CBT) (45 minute sessions for 12 to 16 weeks), augmented by medication treatment when clinically indicated based on the clinical treatment standards. Due to Covid, therapy sessions are offered via remote video conference (in clinic sessions made available if clinically indicated). Cognitive-behavioral therapy (CBT) is a treatment based on learning and cognitive theories. CBT for Obsessive-Compulsive Disorder (OCD) involves gradually exposing patients to anxiety provoking stimuli while having patients refrain from engaging in compulsive rituals and/or avoidance behaviors. There are three major components of CBT treatment for OCD, specifically: (1) exposure to anxiety provoking stimuli, (2) response prevention, and (3) cognitive techniques intended to decrease anxiety during the exposure and response prevention processes.
  Arms: Obsessive Compulsive Disorder
Other: Community Referral as appropriate — Participants with Obsessive Compulsive Symptoms will be referred to the community for treatment
  Arms: Subclinical Obsessive-Compulsive symptoms (OCS)

SUMMARY:
This study will use magnetic resonance imaging (MRI) to assess the function and structure of overlapping task control circuits in children with a range of Obsessive-Compulsive symptoms (OCS). The functioning of task control circuits will be assessed using the well-validated Multisource interference task (MSIT). This study will also assess functional and anatomical connectivity within task control circuits in the same children, and determine whether disturbances in these overlapping circuits are associated with Obsessive-Compulsive Disorder (OCD) symptom severity. Behavioral measures will be administered to further assess regulatory, learning and memory functions. Children with OCD will then be offered a standard course of up to 12 cognitive behavioral therapy (CBT), either via remote video conference sessions or in person visits when clinically indicated, before scanning (along with age-and gender-matched control participants) in order to assess how these circuits may change with treatment. Children with subclinical OC symptoms will be offered referral for treatment on an as-needed basis. In addition, de-identified data may be used in the future to conduct secondary data analyses. As more about OC symptoms and neurobiological mechanisms of interest in the current study are understood, data may be used to answer questions beyond those described in this protocol. All study procedures will be conducted on-site at Columbia University/the New York State Psychiatric Institute (New York, NY) and the University of Michigan's outpatient Child and Adolescent Psychiatry (Ann Arbor, Michigan).

DETAILED DESCRIPTION:
Recruitment is complete. U.S. Department of Health and Human Services OHRP issued an FWA restriction on NYSPI research that included a pause of human subjects research as of June 23, 2023. This study will resume analysis of results from its two sites for results reporting after OHRP and the IRB has approved the resumption of research.

ELIGIBILITY:
Obsessive-Compulsive Disorder (OCD) patient group

INCLUSION:

1. Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) Diagnosis of OCD as the principal problem
2. Not on psychotropic medication and not receiving current psychotherapy for OCD
3. Written informed assent by the participants and consent by the parent
4. Participants and a parent/guardian must be able to read and understand English

EXCLUSION

1. DSM-5 current diagnosis of major depressive disorder, or substance/alcohol abuse
2. DSM-5 lifetime diagnosis of psychotic disorder, bipolar disorder, eating disorder, pervasive developmental disorder, or substance/alcohol abuse
3. Individuals who are currently receiving CBT, other forms of psychotherapy, or psychotropic medications (stable doses of stimulants or other types of ADHD medications - e.g. Guanfacine - are allowable for OCD subjects with comorbid attention deficit hyperactivity disorder following investigator review of medication; on day of study scan, subjects must be willing to refrain from taking medication until after scan is completed)
4. Active suicidal ideation
5. Females who are pregnant or nursing
6. Major medical or neurological problems
7. Presence of metallic device or dental braces
8. Intelligence Quotient (IQ)<80
9. A current or past diagnosis of pediatric autoimmune neuropsychiatric disorders associated with streptococcus (PANDAS)
10. Individuals who are currently receiving CBT, other forms of psychotherapy, or psychotropic medications
11. Individuals who have received a full course of CBT in the past
12. A positive pregnancy test
13. Positive urine screen for illicit drugs

Healthy controls

INCLUSION:

1. Written informed assent by the participants and consent by the parent
2. Participants and a parent/guardian must be able to read and understand English

EXCLUSION:

1. Any current or lifetime psychiatric diagnosis
2. Active suicidal ideation
3. Females who are pregnant or nursing
4. Major medical or neurological problems
5. Presence of metallic device or dental braces
6. IQ <80
7. A current or past diagnosis of pediatric autoimmune neuropsychiatric disorders associated with streptococcus (PANDAS)
8. A positive pregnancy test
9. Positive urine screen for illicit drugs

Obsessive Compulsive Symptoms

INCLUSION:

1. Presence of obsession(s) and/or compulsion(s) but no current diagnosis of OCD (i.e.,<1 hour/day, no more than mild interference or distress)
2. Not on psychotropic medication and not receiving current psychotherapy for OCD
3. Written informed assent by the participants and consent by the parent
4. Participants and a parent/guardian must be able to read and understand English

EXCLUSION:

1. DSM-5 current diagnosis of major depressive disorder, attention-deficit hyperactivity disorder, Tourette's/Tic Disorder, or substance/alcohol abuse
2. DSM-5 lifetime diagnosis of psychotic disorder, bipolar disorder, eating disorder, pervasive developmental disorder, or substance/alcohol abuse
3. Active suicidal ideation
4. Females who are pregnant or nursing
5. Major medical or neurological problems
6. Presence of metallic device or dental braces
7. IQ<80
8. A current or past diagnosis of pediatric autoimmune neuropsychiatric disorders associated with streptococcus (PANDAS)
9. Individuals who are currently receiving CBT, other forms of psychotherapy, or psychotropic medications
10. Individuals who have received a full course of CBT in the past
11. Positive urine screen for illicit drugs

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 169 (Actual)
Dates: Start 2019-03-24 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-06-03 (Actual)

PRIMARY OUTCOMES:
Blood oxygen-level dependent (BOLD) functional MRI signal during a cognitive conflict task | up to 16 weeks after baseline (following 12 weeks of therapy for intervention groups); approximately 15-20 minutes

SECONDARY OUTCOMES:
Blood oxygen-level dependent (BOLD) functional connectivity MRI of task control circuits | up to 16 weeks after baseline (following 12 weeks of therapy for intervention groups);approximately 10 minutes
Child Yale-Brown Obsessive Compulsive Scale | up to 16 weeks after baseline (following 12 weeks of therapy for intervention groups);approximately 1 hour
  Child Yale-Brown Obsessive Compulsive Scale (CYBOCS) is scored on a scale of 0 to 40, with 40 being the most severe.
Obsessive Compulsive Inventory - Child Version (OCI-CV) | baseline assessment of all participants (OCD, subclinical OCS and HC)
  Self-report assessment of obsessive compulsive symptoms, non-clinical to clinical range.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - New York State Psychiatric Institute, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be shared between sites at the University of Michigan and Columbia. A DUA will also be established per University guidelines as required. Coded, de-identified IPD will be shared with the NIMH data repository, RDoCdb.
Supporting Information: SAP, ICF

REFERENCES:
- [Derived] Wang Z, Fontaine M, Cyr M, Rynn MA, Simpson HB, Marsh R, Pagliaccio D. Subcortical shape in pediatric and adult obsessive-compulsive disorder. Depress Anxiety. 2022 Jun;39(6):504-514. doi: 10.1002/da.23261. Epub 2022 Apr 29. PMID 35485920

DOCUMENTS (1):
  • Informed Consent Form (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT03584945/ICF_000.pdf